CLINICAL TRIAL: NCT00662571
Title: A Probe Study of Acamprosate: Genes Associated With Response
Brief Title: Acamprosate: Genes Associated With Response
Acronym: ACAM
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Samuel C. Johnson Foundation (Unknown)
Responsible Party: David Mrazek, M.D., Mayo Clinic
Other Study IDs: 07-007204; P20-acam
Record Dates: First submitted 2008-04-14; First posted 2008-04-21 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Alcoholism
Keywords: nucleotide polymorphisms; disequilibrium haplotype; acamprosate; differentiate; pharmacogenomic; effective individualized treatment; alcohol dependent; N-methyl-D-aspartate receptor (NMDA); metabotropic glutamate receptor; decreasing craving; abstinence maintenance
MeSH Terms: conditions — Alcoholism | interventions — Acamprosate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Samples obtained from study "Developing a DNA Repository for Genomic Studies of Addiction: A Pilot Study"
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: Our hypothesis is that effective acamprosate response in alcohol dependent subjects may be influenced by genetically controlled variation in the functionality of the N-methyl-D-aspartate receptor (NMDA) and/or the type 5 metabotropic glutamate receptor (mGluR5). Hypothesis confirmation could lead to development of effective individualized treatment recommendations for alcohol dependent patients based on pharmacogenomically relevant genetic variations.
  There will be no placebo drug given. Just measurement of genetic response.
  Interventions: Drug: acamprosate

INTERVENTIONS:
Drug: acamprosate — acamprosate 333mg tabs, 2tabs 3times per day = 1998mg/day
  Other Names: Campral is the brand name of acamprosate.

SUMMARY:
In 2004, acamprosate was approved in the U.S. for abstinence maintenance, by decreasing craving, in alcoholic patients who have undergone detoxification. while a new anti-craving drug was encouraging, only 36.1% of the subjects treated with acamprosate remained abstinent for 6 months. Having the ability to identify treatment responsive individuals would have a major impact on the use of acamprosate.

DETAILED DESCRIPTION:
The primary objective of this pharmacogenomic probe study of acamprosate is to identify genetic variations that predict response. Our hypothesis is that effective acamprosate response in alcohol dependent subjects may be influenced by genetically controlled variation in the functionality of the N-methyl-D-aspartate receptor (NMDA) and/or the type 5 metabotropic glutamate receptor (mGluR5). Hypothesis confirmation could lead to development of effective individualized treatment recommendations for alcohol dependent patients based on pharmacogenomically relevant genetic variations.

The general goal is to identify genetic polymorphic variants that differentiate subjects continuously abstinent for six months while taking acamprosate from relapsed subjects. The initial analysis will determine whether any of ten polymorphisms in four target genes (GRIN1, GRIN2A and GRIN2B that code for the NMDA receptor and GRM5 that codes for the type mGluR5 receptor) are associated with successful abstinence. Subsequent analyses will examine whether variation in a comprehensive set of 383 linkage disequilibrium haplotype tagged single nucleotide polymorphisms of these four genes predicts successfully abstinent subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females, Age 18-80.
2. 2. Primary diagnosis of alcohol dependence based on DSM-IV-TR criteria and determined by the Psychiatric Research Interview for Substance and Mental Disorders (PRISM) (stable mood and anxiety disorders will not be exclusionary).
3. Prior enrollment in the IRB approved protocol "Developing a DNA Repository for Genomic Studies of Addiction: A Pilot Study".

Exclusion Criteria:

1. Inability to provide informed consent.
2. Inability to speak English.
3. History of hypersensitivity or allergic reaction to acamprosate.
4. Moderate to severe renal impairment, as determined by a creatinine level > 1.5 mg/dL.
5. Diagnosis of primary biliary cirrhosis, chronic active hepatitis, and drug-induced hepatic insufficiency, as noted in the medical record.
6. Women who are pregnant, lactating, or are planning to become pregnant during the next year.
7. Any unstable active medical or additional psychiatric condition as determined by the investigator.

9. Active suicidal ideation as determined by responses provided during PRISM or as determined by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects selected from Mayo Clinics Addiction programs.
Sampling Method: Non-Probability Sample
Enrollment: 485 (Actual)
Dates: Start 2008-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Aim 1: To determine the relationship between genetically determined variation in the NMDA receptor and treatment response to acamprosate. | 6 months

SECONDARY OUTCOMES:
Aim 2: To determine the relationship between genetically determined variation in the mGluR5 receptor and treatment response to acamprosate. | 6months

CONTACTS AND LOCATIONS:
Overall Officials: David Mrazek, M.D., Principal Investigator — Mayo Clinic, Department of Psychiatry
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Ho MF, Zhang C, Cohan JS, Tuncturk M, Heider RM, Coombes BJ, Biernacka J, Moon I, Skime M, Ho AM, Ngo Q, Skillon C, Croarkin PE, Oesterle TS, Karpyak VM, Li H, Weinshilboum RM. IL17RB genetic variants are associated with acamprosate treatment response in patients with alcohol use disorder: A proteomics-informed genomics study. Brain Behav Immun. 2024 Aug;120:304-314. doi: 10.1016/j.bbi.2024.06.007. Epub 2024 Jun 8. PMID 38852760
- [Derived] Ho MF, Zhang C, Moon I, Biernacka J, Coombes B, Ngo Q, Skillon C, Skime M, Oesterle T, Croarkin PE, Karpyak VM, Li H, Weinshilboum RM. Epigenetic regulation of GABA catabolism in iPSC-derived neurons: The molecular links between FGF21 and histone methylation. Mol Metab. 2023 Nov;77:101798. doi: 10.1016/j.molmet.2023.101798. Epub 2023 Sep 7. PMID 37689244
- [Derived] Karpyak VM, Coombes BJ, Geske JR, Pazdernik VM, Schneekloth T, Kolla BP, Oesterle T, Loukianova LL, Skime MK, Ho AM, Ngo Q, Skillon C, Ho MF, Weinshilboum R, Biernacka JM. Genetic predisposition to major depressive disorder differentially impacts alcohol consumption and high-risk drinking situations in men and women with alcohol use disorder. Drug Alcohol Depend. 2023 Feb 1;243:109753. doi: 10.1016/j.drugalcdep.2022.109753. Epub 2022 Dec 24. PMID 36608483
- [Derived] Ho MF, Zhang C, Moon I, Wei L, Coombes B, Biernacka J, Skime M, Choi DS, Frye M, Schmidt K, Gliske K, Braughton J, Ngo Q, Skillon C, Seppala M, Oesterle T, Karpyak V, Li H, Weinshilboum R. Genome-wide association study for circulating FGF21 in patients with alcohol use disorder: Molecular links between the SNHG16 locus and catecholamine metabolism. Mol Metab. 2022 Sep;63:101534. doi: 10.1016/j.molmet.2022.101534. Epub 2022 Jun 22. PMID 35752286
- [Derived] Karpyak VM, Biernacka JM, Geske JR, Abulseoud OA, Brunner MD, Chauhan M, Hall-Flavin DK, Lewis KA, Loukianova LL, Melnyk GJ, Onsrud DA, Proctor BD, Schneekloth TD, Skime MK, Wittkopp JE, Frye MA, Mrazek DA. Gender-specific effects of comorbid depression and anxiety on the propensity to drink in negative emotional states. Addiction. 2016 Aug;111(8):1366-75. doi: 10.1111/add.13386. Epub 2016 May 5. PMID 27009547